CLINICAL TRIAL: NCT04386434
Title: Active for Life Assisted Living Feasibility and Acceptability Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic, researchers no longer have access to residents of assisted living.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Janet L. Larson, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00175558
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Sedentary Behavior
Keywords: assisted living; physical activity; sedentary behavior; self-efficacy
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active for Life (Experimental): The Active Life intervention includes structured walking, functional circuit training, stretching and behavior/educational components.
  Interventions: Behavioral: Active for Life: Assisted Living

INTERVENTIONS:
Behavioral: Active for Life: Assisted Living — Each intervention session will take place within the assisted living facility twice a week for 12 weeks.
  Sessions will begin with 5-10 minutes of walking in the hallway. Participants will be encouraged to walk at their own pace and allowed to take breaks if needed.
  Next, behavioral strategies based on the construct of self-efficacy from social cognitive theory and education about physical activity will be delivered. This component is scheduled between the walking and circuit training, lasts 15-20 minutes, and serves as a rest period.
  Circuit training will focus on strength and balance. Approximately 8 exercise stations will be set up, and the exercises performed at each station will be changed approximately every 4 weeks. The circuit training will last ~30-40 minutes, with participants moving from one station to the next at their own pace and taking breaks in between.

SUMMARY:
This study examines the effects of a physical activity and behavioral program, called Active for Life, to promote increased physical activity and reduced sedentary behavior of older adults who live in assisted living. A sedentary lifestyle is very common in this population and if this program is successful it will be used to promote physical activity and improve the health of older adults in assisted living.

DETAILED DESCRIPTION:
Sedentary behavior (SB) is an emerging health risk, especially for older adults, as it is associated with chronic disease, loss of function, and increased disability and frailty. Older adults in assisted living (AL) are less active than their peers living independently. Recent evidence demonstrates there are substantial health benefits from light physical activity (LPA) and the newly published Physical Activity Guidelines for Americans recommends that older adults replace SB with LPA. An intervention to increase LPA and reduce SB has potential to reduce health risks, slow functional decline and frailty, and delay residents' needs for higher-level care such as a nursing home. We propose to test the feasibility and acceptability of a self-efficacy based intervention, "Active for Life," with the goal of increasing PA and decreasing SB of AL residents.

Active for Life is a 12 week intervention. Key components include (a) exercise with functional circuit training (FCT), walking, and stretching, (b) a behavioral component with a structured self-efficacy enhancing intervention that includes self-regulation strategies, and (c) education that addresses principles of exercise, the distinct health benefits of LPA, the negative consequences of too much sedentary time, and strategies for overcoming barriers to physical activity. It is important to test the feasibility and acceptability of the intervention for AL residents because this population will be more frail than previously tested populations. The intervention has been modified to be appropriate for AL residents based on guidance from AL experts and individual interviews conducted with AL residents. We will enroll 27 participants from approximately four AL facilities. Outcomes will be measured at baseline and at conclusion of the intervention. The primary outcomes are feasibility and acceptability of the intervention, but we will also examine preliminary evidence of outcome measures of objectively-measured sedentary behavior and physical activity, self-efficacy for exercise, value of physical activity, self-rated health, physical function, anxiety, depression, pain interference, and fatigue. This study is innovative because there are no well-established evidence-based interventions to promote PA in the AL setting and none that focus on increasing LPA and decreasing SB.

ELIGIBILITY:
Inclusion Criteria:

* Residing in assisted living facility
* Inactive (performing moderate level activities for less than 30 min./day, 5 day/week or not performing muscle strengthening activities twice/week) or a desire to increase physical activity
* Score of at least 3 on the Mini-Cog cognitive screening

Exclusion Criteria:

* Mobility issues that prevent participation in PA, such as if they rely on a wheelchair or motorized scooter (not excluded if they require an assistive device such as a cane or walker)
* Hospitalization in the previous month
* Skin on the thigh where ActivPAL monitor would be placed is not intact (has lesions, signs of infection, rash, or skin breakdown)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Number of participants screened | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate how many participants volunteered to be screened for participation in the study.
Feasibility: Number of participants eligible | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate how many participants met eligibility criteria for study participation.
Feasibility: Numbers of participants ineligible by each eligibility criterion | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will summarize reasons that participants were ineligible for study participation by adding up the number of people who don't meet each specific eligibility criterion.
Feasibility: Number of participants who enroll | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate how many eligible participants decide to enroll in the study.
Feasibility: Length of time for recruitment activities | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate how much time is spent to recruit the study sample.
Feasibility: Percentage of activity sessions attended by participants | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate the percentage of activity sessions that participants attended.
Feasibility: Participant retention rates | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will calculate retention rates of how many participants started and how many completed the study.
Feasibility: Documentation of stated reasons for participant dropout | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will document stated reasons for dropout from the study as much as we are able.
Feasibility: Injuries and adverse events | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will summarize any adverse events/injuries that occur during the study.
Feasibility: Rates of missing or unusable data | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will summarize how much data are missing from baseline, mid-intervention, and post-intervention data collections.
Feasibility: Time required to complete outcome measures | After completion of the 12 week intervention
  Several measures will be used to describe the feasibility of the intervention. We will keep record of how long each data collection session takes and calculate average length of data collection at both baseline and post-intervention.
Acceptability: Exit interviews | After completion of the 12 week intervention
  Semi-structured exit interviews will ask questions related to acceptability of the intervention, such as how participants felt about the overall intervention and its specific components, whether the time commitment was reasonable, whether assisted living staff were supportive of their participation and goals, and any suggestions for future improvements.
Acceptability: Final acceptability scale | After completion of the 12 week intervention
  This scale consists of 13 questions related to participants' overall satisfaction with the intervention and its components. Higher score indicates greater intervention acceptability.

SECONDARY OUTCOMES:
Time spent in sedentary behavior and physical activity | 7 days of data are gathered at baseline at after the 12 week intervention.
  ActivPAL monitor will measure time spent sitting/lying, standing, and stepping for 7 consecutive days at each measurement.
Self-efficacy for exercise | Measured at baseline, three weeks, and after 12 week intervention.
  Exercise self-efficacy- 9 items. Potential range of scores is 0 to 90. Higher score indicates higher self-efficacy for exercise.
Value of Physical Activity | Measured at baseline and after 12 week intervention.
  Single item asking "How important is physical activity in your life?" with a Likert response scale ranging from 1 to 5. Higher score will indicate greater importance of physical activity
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health | Measured at baseline and after 12 week intervention.
  Physical, social, and mental health- 10 items. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low global health and higher scores indicate higher global health.
PROMIS Physical Functioning | Measured at baseline and after 12 week intervention.
  Physical function scale- measured with computer adaptive testing. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low physical function and higher scores indicate higher physical function.
PROMIS Anxiety | Measured at baseline and after 12 week intervention.
  General experience with anxious moods- measured with computer adaptive testing. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low anxiety and higher scores indicate higher anxiety.
PROMIS Depression | Measured at baseline and after 12 week intervention.
  General experience with depressed moods- measured with computer adaptive testing. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low depression and higher scores indicate higher depression.
PROMIS Fatigue | Measured at baseline and after 12 week intervention.
  General experience of fatigue- measured with computer adaptive testing. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low fatigue and higher scores indicate higher fatigue.
PROMIS Pain Interference | Measured at baseline and after 12 week intervention.
  Extent to which pain interferes with functioning- measured with computer adaptive testing. Scores are calculated as T-scores with a mean = 50 and standard deviation = 10. Low scores indicate low pain interference and higher scores indicate higher pain interference.
Positive and Negative Social Influences on PA in Older Adults | Measured at baseline and after 12 week intervention.
  Support from family and friends for being physically active. The questionnaire has 27 items (15 items describing positive social influence and 12 items describing negative social influence). The potential range of scores for positive social influence is 0 to 180 and the potential range of scores for negative social influence is 0 to 144.
Acceptability: Mid-point acceptability scale | Measured at 6-weeks (mid-point of intervention)
  This scale consists of 3 questions related to acceptability of intervention delivery. Higher score indicates greater intervention acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Larson, PhD, RN, Principal Investigator — University of Michigan School of Nursing
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
At this point the investigators have no plans to share IPD, but would consider a request to share deidentified data if it had the potential to advance science in the promotion of physical activity for older adults